CLINICAL TRIAL: NCT01397344
Title: Patients' Preferences for Traditional Medicine Doctor's Attire
Status: Completed | Type: Observational
Sponsor: Korean Medicine Hospital of Pusan National University (Other)
Responsible Party: Principal Investigator, Jun-Yong Choi, Associate professor, Korean Medicine Hospital of Pusan National University
Other Study IDs: KCRC-IRB-2011008
Record Dates: First submitted 2011-07-14; First posted 2011-07-19 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Attire Preference
Keywords: People in the outpatient waiting room

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Doctors' attire has known to impact patients' trust and confidence for better clinical practice. However, few survey research regarding this topic has been conducted in traditional asian medicine field. The aim of our study is to determine whether traditional medicine doctor's attire impacts on patients' confidence and trust.

Participants will be given randomly one set of photographs from the 2 kind of photographs, i.e., photographs of a male or female doctor, each set dressed in 4 different styles.

After this, they will be asked to report their preferences for the 4 styles of dress according to given questions and they will answer the degree of their feeling on the importance of Korean Medicine doctor's appearance.

DETAILED DESCRIPTION:
After seeing one set of photographs, participants will answer the questions below.

Choose the most appropriate attire from the four dressing styles (a.formal wear b.conventional white coat c.white coat in traditional form d. casual wear) to the questions below (1-10).

1. Which attire of Korean medicine doctor would you trust the most?
2. Which attire of Korean medicine doctor would you be more likely to follow their advice?
3. Which attire of Korean medicine doctor would you recommend to your acquaintance?
4. Which attire of Korean medicine doctor would you be the most comfortable ?
5. Which attire of Korean medicine doctor would you prefer to discuss an intimate social problem or a private issue?
6. Which attire of Korean medicine doctor would you prefer for a minor medical problem(eg, a cold)?
7. Which attire of Korean medicine doctor would you expect to be the most clean?
8. Which attire of Korean medicine doctor would you expect to be the most hygienic?
9. Which attire of Korean medicine doctor would you expect not to spread infectious germs to others?
10. Which attire of Korean medicine doctor would you have the most confidence in their diagnosis and treatment when they perform clinical examination by touching you?
11. How strongly do you feel about the importance of Korean medicine doctor's appearance?

    1. extremely important
    2. quite important
    3. important
    4. a little important
    5. not at all important

ELIGIBILITY:
Inclusion Criteria:

* More than 19 years old, less than 80 years old at the time of the study
* Outpatients from diverse clinic departments in Korean Medicine Hospital of Pusan National University, Yangsan, Korea

Exclusion Criteria:

* Subjects who are demented, noncommunicative, or blind
* Companion(s) of the interviewee

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People in the Outpatient Waiting Room
Sampling Method: Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2011-07; Primary Completion 2012-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Patient's preference for a specific attire of the traditional medicine doctor from four different styles of dress. | During day one visit (lasting an average of 1-3 hours)
  Patients will choose the most appropriate attire from four dressing styles (formal suit, conventional white coat, white coat in traditional form and casual wear).

SECONDARY OUTCOMES:
Participants' feeling about the importance of Korean Medicine doctor's appearance. | During day one visit (lasting an average of 1-3 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Yong Choi, MS, Principal Investigator — Korean Medicine Hospital of Pusan National University
Locations (1):
- Korean Medicine Hospital of Pusan National University, Yangsan, Gyeongsangnam-do, South Korea